CLINICAL TRIAL: NCT05586425
Title: Neuroplastic Adaptations in Youth at High Risk for Developing Psychopathology: A Randomized Controlled Trial Modelling Feasibility and Clinical Improvement Following ERS Training With Changes in Brain Connectivity and Anatomy
Brief Title: Neuroplastic Adaptations in Youth at High Risk for Developing Psychopathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13517
Record Dates: First submitted 2022-07-21; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Emotion Regulation
Keywords: Neuroplastic Adaptations; Psychopathology
MeSH Terms: conditions — Emotional Regulation | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotion Regulation Skills + Treatment as Usual (Experimental): Emotion Regulation Skills (ERS), a version of Dialectical Behaviour Therapy Skills Training, is a type of skills-focused therapy for individuals who experience severe emotion dysregulation.
  Interventions: Behavioral: Emotion Regulation Skills + Treatment as Usual
- Treatment as Usual (Active Comparator): Treatment as Usual entails psychiatric medication management, psychiatric management, individual support from peer mentors, drop-in activity groups, etc.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Emotion Regulation Skills + Treatment as Usual — ERS has been updated to be friendlier to youth and involves learning skills for how to: (1) be more present in the moment, (2) effectively manage and respond to emotional experiences, (3) communicate your needs to others, and (4) increase your ability to tolerate distress.
  Arms: Emotion Regulation Skills + Treatment as Usual
Behavioral: Treatment as Usual — Treatment as Usual entails psychiatric medication management, psychiatric management, individual support from peer mentors, drop-in activity groups, etc.
  Arms: Treatment as Usual

SUMMARY:
This pilot study aims to inform decision-making for a bigger study we intend to conduct in the future. The larger investigation will explore how helpful a treatment program for youth (ages 17 - 24) with emotion dysregulation (ED) is, as well as how this program affects the brain. The current pilot study will also explore these topics, but on smaller scale.The treatment program we are researching is called Emotion Regulation Skills (ERS). It is based on Dialectical Behaviour Therapy Skills Training (DBT-ST), a type of skills-focused therapy for individuals who experience severe ED. ERS has been updated to be friendlier to youth and involves learning skills for how to: (1) be more present in the moment, (2) effectively manage and respond to emotional experiences, (3) communicate your needs to others, and (4) increase your ability to tolerate distress.

DETAILED DESCRIPTION:
Emotion dysregulation (ED), described as an individual's inability to respond to and cope with their emotions, has been linked to many serious mental health problems, including substance use and suicide. Minority stress, defined as the additional stress that members of marginalized groups experience because of the prejudice and discrimination they face, is also believed to be linked with ED. Youth are particularly prone to developing ED. As such, it is important to offer evidence-based treatment interventions to this age group in order to offset problems associated with ED and promote mental wellness in adulthood. Dialectical Behaviour Therapy Skills Training (DBT-ST) is proven to be an effective intervention for reducing ED in youth. This pilot study will offer a 14-week, youth-friendly version of DBT-ST, called Emotion Regulation Skills (ERS), to youth with ED. Half of the participants in this study will complete ERS in the Youth Wellness Centre (YWC) at St. Joseph's Healthcare Hamilton (SJHH), in addition to receiving all interventions typically associated with treatment as usual (TAU). The other half will be placed on a waitlist for ERS, and will only receive TAU for 14 weeks. After 14 weeks, the TAU group will be crossed over into the intervention condition, at which point they will also receive ERS. The primary purpose of this pilot study will be to assess the feasibility of a larger study to measure clinical improvement in youth who participate in ERS. As secondary objectives, this pilot study will also collect data on clinical and brain-based outcomes following ERS. For this study, all participants will be asked to undergo fMRI neuroimaging and respond to specific questionnaires about their levels of ED and other mental health symptoms before and after 14 weeks of ERS or TAU. Participants in the TAU group will undergo a third session of fMRI neuroimaging and respond to questionnaires after they have also completed ERS, 14 weeks after being crossed over into the intervention condition (i.e., 28 weeks after their first neuroimaging/questionnaires). It is expected that ERS will improve ED more than TAU after 14 weeks, and that these changes will be evident at the brain level. It is also expected that these changes will be greater in cisgender individuals than in transgender and gender diverse (TGD) individuals, who are at greater risk for experiencing minority stress related to their gender identity.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 17 and 24 years, inclusive
* Difficulties in Emotion Regulation Scale score >96 at baseline
* Able to provide written informed consent and communicate in English

Exclusion Criteria:

* Diagnosis of an active substance use disorder (SUD)
* Diagnosis of an organic brain disorder
* Lifetime history of a psychotic disorder (e.g., bipolar affective disorder, schizophrenia, schizoaffective disorder, etc.)
* Active PTSD symptoms
* Currently using antidepressants, only if the last adjustment in dose was within 3 months of beginning the study
* Has received standard DBT treatment in the past 2 years
* MRI contraindications

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate (Feasibility Threshold) | 14 weeks
  Assessed by the total number of participants recruited from one site during the recruitment period
  (i.e., Is one site sufficient for recruitment or will the larger study require additional sites or strategies to recruit the necessary sample size? Is it plausible to recruit the required number of TGD individuals?)
Eligibility Participants (Feasibility Threshold) | 14 weeks
  Assessed by changes in the baseline number of participants contacted to the number of failed screening assessments
  (i.e., Are the criteria too narrow? What is the rate of individuals being contacted to participate in the study, but failing screening assessments?)
Length of Completion of Procedures (Feasibility Threshold) | 14 weeks
  Assessed by comparing the actual time required per session to the anticipated 3-hour allotment for assessments
  (i.e., Is the actual time required per study visit different from what is anticipated?)
Location Logistics (Feasibility Threshold) | 14 weeks
  Assessed by subjective evaluation and feedback from the research assistant
  (i.e., Are there unforeseen difficulties due to the Imaging Research Centre being located in a different place than the YWC?)
Attrition Rate (Feasibility Threshold) | 14 weeks
  Assessed by changes from the baseline number of participants to those retained at 14 weeks (i.e., What percentage of individuals drop out of ERS and the study?)
Intervention Attendance Rates (Feasibility Threshold) | 14 weeks
  Assessed by comparing the number of sessions attended to the total number of sessions allocated (i.e., On average, how many ERS sessions do individuals attend?)
Burdensomeness of Study Procedures (Feasibility Threshold) | 14 weeks
  Assessed by subjective evaluation provided by study participants
  (i.e., Are study procedures too lengthy or onerous for participants?)
Research Impact on the Youth Wellness Centre (YWC) | 14 weeks
  Assessed by a subjective review and feedback from the clinical team, up to 14 weeks
  (i.e., How do YWC staff perceive the impact of research procedures on their own logistics?)
Communication between Clinical and Research staff | 14 weeks
  assessed by subjective review and feedback from the clinical team, up to 14 weeks

SECONDARY OUTCOMES:
Emotion Dysregulation and other relevant symptoms/conditions | 14 weeks
  Changes in the Difficulties in Emotion Regulation Scale (DERS) from baseline to 14 weeks; compared within (pre and post) and between groups (ERS and TAU)
  The DERS is a 36-item, self-report measure of emotion dysregulation with a 5-point Likert scale (1 = "almost never" to 5 = "almost always). Improvement of 20% or greater on the DERS will be considered significant clinical improvement.
Resting-state functional connectivity (rs-FC) | 14 weeks
  Changes in blood-oxygen-level-dependent (BOLD) signal (measured by fMRI) from baseline to 14 weeks; compared within (pre and post) and between groups (ERS and TAU)
Emotion Dysregulation and brain connectivity between limbic and prefrontal brain areas | 14 weeks
  Changes in the DERS scale compared to changes in blood-oxygen-level-dependent (BOLD) signal (measured by fMRI) in the limbic and prefrontal brain regions from baseline to 14 weeks; compared within (pre and post) and between groups (ERS and TAU)

CONTACTS AND LOCATIONS:
Overall Officials: Maiko Schneider, MD/PhD, Principal Investigator — McMaster University

REFERENCES:
- [Background] O'Neill A, D'Souza A, Samson AC, Carballedo A, Kerskens C, Frodl T. Dysregulation between emotion and theory of mind networks in borderline personality disorder. Psychiatry Res. 2015 Jan 30;231(1):25-32. doi: 10.1016/j.pscychresns.2014.11.002. Epub 2014 Nov 13. PMID 25482858
- [Background] Gratz KL, Moore KE, Tull MT. The role of emotion dysregulation in the presence, associated difficulties, and treatment of borderline personality disorder. Personal Disord. 2016 Oct;7(4):344-353. doi: 10.1037/per0000198. PMID 27709991